CLINICAL TRIAL: NCT01591785
Title: An Investigator-Initiated Study: Treatment of Staphylococcus Aureus Colonization in Hand Eczema Decreases Severity of Disease
Brief Title: Treatment of Staphylococcus Aureus Colonization in Hand Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Goldenberg (Other)
Responsible Party: Sponsor-Investigator, Gary Goldenberg, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 11-0038
Record Dates: First submitted 2012-04-30; First posted 2012-05-04 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Hand Eczema; Foot Eczema
Keywords: Hand; Foot; Eczema; Atopic Dermatitis
MeSH Terms: conditions — Eczema; Dermatitis, Atopic | interventions — retapamulin; Ointments; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retapamulin 1% ointment (Active Comparator): Retapamulin 1% ointment for 5 days AND clobetasol propionate foam for 14 days
  Interventions: Drug: Retapamulin 1% ointment
- Placebo ointment (Placebo Comparator): Placebo ointment for 5 days AND clobetasol propionate foam for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retapamulin 1% ointment — Retapamulin 1% ointment for 5 days AND clobetasol propionate foam for 14 days
  Other Names: Altabax and Olux Foam
  Arms: Retapamulin 1% ointment
Drug: Placebo — Placebo ointment for 5 days AND clobetasol propionate foam for 14 days
  Other Names: Petroleum jelly
  Arms: Placebo ointment

SUMMARY:
Atopic dermatitis is a chronic disease characterized by itching and eczematous lesions. In adults, eczema commonly localizes to the hands or feet. Several studies have implicated bacterial contamination, especially with Staphylococcus aureus (S. aureus), to be a factor in atopic dermatitis, as infection with this bacteria correlates with disease severity. No trial to date has investigated how to treat S. aureus infection in adults with hand or hand/foot dermatitis. Using retapamulin ointment in the nose and on the hands or hands/feet, the investigators expect to have a significant clearance rate of s. aureus infection. The investigators believe that treating the bacterial infection along with treating the condition with a topical corticosteroid will significantly decrease the severity of hand/foot dermatitis in our study population.

DETAILED DESCRIPTION:
Primary Study Objectives:

1. To evaluate the efficacy of retapamulin 1% ointment with clobetasol propionate 0.05% foam versus vehicle ointment with clobetasol propionate 0.05% foam as a treatment regimen for hand or hand/foot atopic dermatitis.
2. To evaluate the incidence of intranasal and hand/foot S aureus carriage rates in subjects with hand/foot atopic dermatitis via cultures of an anterior nare and the most severely graded target lesion of the hand/foot dermatitis.
3. To evaluate the incidence of mupirocin-resistance and methicillin-resistance in S aureus isolates in subjects with hand/foot atopic dermatitis via cultures of an anterior nare and the most severely graded target lesion of the hand/foot dermatitis.

Primary and secondary endpoints will be analyzed by appropriate statistical models by a qualified statistician. Any results of this pilot study will be treated as exploratory and hypothesis generating.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age with a clear diagnosis of moderate-to-severe hand or hand/foot dermatitis.
* Subjects must be in general good health as confirmed by a medical history.
* Subjects must be capable of understanding and willing to provide a signed and dated written voluntary informed consent before any protocol specific procedures are performed.
* At the Baseline Visit, Subjects must have a Physician's Global Assessment (PGA) of at least 3 (moderate severity).
* Subject must be willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up period periods and comply with all study requirements.
* If a subject is a female of childbearing potential she must have a negative urine pregnancy test prior to study treatment initiation and must agree to use an approved method of birth control during the study period (barrier, oral, injection, intrauterine). NOTE: Post-menopausal (amenorrhea for at least one year) or surgically sterile (tubal ligation and/or hysterectomy) females are categorized as non-childbearing potential.

Exclusion Criteria:

* Non-English speaking subjects
* Females who are pregnant, breast feeding, or attempting to conceive.
* Subjects with a history of known or suspected intolerance to any of the excipients of retapamulin 1% ointment or clobetasol propionate 0.05% foam.
* Subjects who have used any topical corticosteroids, topical antibiotics, topical immunosuppressants, other topical therapies (tar, calcineurin inhibitors), or phototherapy (PUVA, UVB) within eight weeks of the Baseline Visit.
* Subjects who have used any systemic corticosteroids, systemic antibiotics, or systemic immunosuppressants therapies within eight weeks of the Baseline Visit.
* Subjects with any overt signs of skin atrophy, telangiectasias, and/or striae in the target area(s).
* Subjects with any active skin malignancy.
* Subjects requiring the use of medications known to alter the course of atopic dermatitis during the study period.
* Subjects who are currently participating in or, within the previous 28 days, have participated in another study for the treatment for atopic dermatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Goldenberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Meding B, Lantto R, Lindahl G, Wrangsjo K, Bengtsson B. Occupational skin disease in Sweden--a 12-year follow-up. Contact Dermatitis. 2005 Dec;53(6):308-13. doi: 10.1111/j.0105-1873.2005.00731.x. PMID 16364116
- [Background] Williams RE, Gibson AG, Aitchison TC, Lever R, Mackie RM. Assessment of a contact-plate sampling technique and subsequent quantitative bacterial studies in atopic dermatitis. Br J Dermatol. 1990 Oct;123(4):493-501. doi: 10.1111/j.1365-2133.1990.tb01455.x. PMID 2095181
- [Background] Hanifin JM, Rogge JL. Staphylococcal infections in patients with atopic dermatitis. Arch Dermatol. 1977 Oct;113(10):1383-6. PMID 911165
- [Background] Leyden JJ, Marples RR, Kligman AM. Staphylococcus aureus in the lesions of atopic dermatitis. Br J Dermatol. 1974 May;90(5):525-30. doi: 10.1111/j.1365-2133.1974.tb06447.x. No abstract available. PMID 4601016
- [Background] Jensen JM, Folster-Holst R, Baranowsky A, Schunck M, Winoto-Morbach S, Neumann C, Schutze S, Proksch E. Impaired sphingomyelinase activity and epidermal differentiation in atopic dermatitis. J Invest Dermatol. 2004 Jun;122(6):1423-31. doi: 10.1111/j.0022-202X.2004.22621.x. PMID 15175033
- [Background] Arikawa J, Ishibashi M, Kawashima M, Takagi Y, Ichikawa Y, Imokawa G. Decreased levels of sphingosine, a natural antimicrobial agent, may be associated with vulnerability of the stratum corneum from patients with atopic dermatitis to colonization by Staphylococcus aureus. J Invest Dermatol. 2002 Aug;119(2):433-9. doi: 10.1046/j.1523-1747.2002.01846.x. PMID 12190867
- [Background] Komatsu N, Saijoh K, Kuk C, Liu AC, Khan S, Shirasaki F, Takehara K, Diamandis EP. Human tissue kallikrein expression in the stratum corneum and serum of atopic dermatitis patients. Exp Dermatol. 2007 Jun;16(6):513-9. doi: 10.1111/j.1600-0625.2007.00562.x. PMID 17518992
- [Background] Sandilands A, Terron-Kwiatkowski A, Hull PR, O'Regan GM, Clayton TH, Watson RM, Carrick T, Evans AT, Liao H, Zhao Y, Campbell LE, Schmuth M, Gruber R, Janecke AR, Elias PM, van Steensel MA, Nagtzaam I, van Geel M, Steijlen PM, Munro CS, Bradley DG, Palmer CN, Smith FJ, McLean WH, Irvine AD. Comprehensive analysis of the gene encoding filaggrin uncovers prevalent and rare mutations in ichthyosis vulgaris and atopic eczema. Nat Genet. 2007 May;39(5):650-4. doi: 10.1038/ng2020. Epub 2007 Apr 8. PMID 17417636
- [Background] Haslund P, Bangsgaard N, Jarlov JO, Skov L, Skov R, Agner T. Staphylococcus aureus and hand eczema severity. Br J Dermatol. 2009 Oct;161(4):772-7. doi: 10.1111/j.1365-2133.2009.09353.x. Epub 2009 Jul 3. PMID 19575755
- [Background] Huang JT, Abrams M, Tlougan B, Rademaker A, Paller AS. Treatment of Staphylococcus aureus colonization in atopic dermatitis decreases disease severity. Pediatrics. 2009 May;123(5):e808-14. doi: 10.1542/peds.2008-2217. PMID 19403473
- [Background] Naderer OJ, A.M., Roberts K, et al. , Nasal Decolonization of persistent Staphylococcus aureus carriers with twice daily application of retapamulin ointment, 1%, for 3 or 5 days. , in Presented at the joint 48th annual interscience conference on antimicrobial agents adn chemotherapy at the 46th Annual Meeting of Infectious Diseases Society of America. 2008: Washington DC.
- [Result] Haddican M, Linkner RV, Singer G, Jim SC, Gagliotti M, Goldenberg G. Retapamulin 1% Ointment and Clobetasol Propionate 0.05% Foam is More Efficacious than Vehicle Ointment and Clobetasol 0.05% Propionate Foam in the Treatment of Hand/Foot Dermatitis: A Single Center, Randomized, Double-blind Study. J Clin Aesthet Dermatol. 2014 Jul;7(7):32-6. PMID 25053981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from January 2012 to August 2012, all subjects were enrolled at one site.
Groups:
- Retapamulin 1% Ointment: twice daily topical application of clobetasol propionate foam 0.05% for 14 days and Retapamulin 1% ointment for 5 days
- Placebo Ointment: twice daily topical application of clobetasol propionate foam 0.05% for 14 days and placebo ointment for 5 days
Period: Overall Study
Arm/Group | Retapamulin 1% Ointment | Placebo Ointment
Started | 30 | 30
Completed | 26 | 28
Not Completed | 4 | 2
Not completed — worsening condition | 1 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retapamulin 1% Ointment | Placebo Ointment | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Full Range); unit: years] | 41.5 [22 to 77] | 44.4 [23 to 70] | 43 [22 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 16
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 17 | 23 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Physician Global Assessment (PGA) [Mean (Full Range); unit: units on a scale] — 0 = Clear (no inflammatory signs of atopic dermatitis)
  1. = Almost clear (just perceptible erythema and papulation/infiltration)
  2. = Mild (mild erythema and papulation/infiltration)
  3. = Moderate (moderate erythema and papulation/infiltration, +/- lichenification, +/- excoriation)
  4. = Severe (severe erythema and papulation infiltration, + lichenification/excoriation, +/- oozing/weeping)
  5. = Very severe (very severe erythema and papulation/infiltration, + lichenification, + excoriation, +oozing/weeping)
  units on a scale | 3.5 [3 to 5] | 3.7 [3 to 5] | 3.6 [3 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PGA of 0 or 1
Description: Physician's Global Assessment PGA 0 = Clear (no inflammatory signs of atopic dermatitis)
  1 = Almost clear (just perceptible erythema and papulation/infiltration)
Time Frame: Day 15
Measure: Number; unit: participants
Arm/Group | Retapamulin 1% Ointment | Placebo Ointment
Number analyzed (Participants) | 30 | 30
participants | 22 | 14
Statistical Analysis 1: Comparison: Retapamulin 1% Ointment vs Placebo Ointment; Test type: Superiority or Other; p = 0.035, Chi-squared

2. Primary Outcome: Number of Participants With PGA of 0 or 1
Description: as for outcome 1
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | Retapamulin 1% Ointment | Placebo Ointment
Number analyzed (Participants) | 30 | 30
participants | 15 | 11
Statistical Analysis 1: Comparison: Retapamulin 1% Ointment vs Placebo Ointment; Test type: Superiority or Other; p = 0.28, Chi-squared

3. Secondary Outcome: Staph Aureus Culture Results
Description: The percentage of subjects who had both negative S. aureus skin and nares cultures with a PGA of clear/almost clear at day 15 compared to baseline
Time Frame: Day 15
Measure: Number; unit: percentage of participants
Arm/Group | Retapamulin 1% Ointment | Placebo Ointment
Number analyzed (Participants) | 30 | 30
percentage of participants | 61 | 30
Statistical Analysis 1: Comparison: Retapamulin 1% Ointment vs Placebo Ointment; Test type: Superiority or Other; p = 0.0495, Chi-squared

4. Secondary Outcome: Staph Aureus Culture Results
Description: The percentage of subjects who had both negative S. aureus skin and nares cultures with a PGA of clear/almost clear at day 28 compared to baseline
Time Frame: Day 28
Measure: Number; unit: percentage of participants
Arm/Group | Retapamulin 1% Ointment | Placebo Ointment
Number analyzed (Participants) | 30 | 30
percentage of participants | 28 | 13
Statistical Analysis 1: Comparison: Retapamulin 1% Ointment vs Placebo Ointment; Test type: Superiority or Other; p = 0.27, Chi-squared

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Retapamulin 1% Ointment | Placebo Ointment
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retapamulin 1% Ointment (N=30) | Placebo Ointment (N=30)
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Eczema flare (Skin and subcutaneous tissue disorders) | 1 | 1
Dryness (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study size was small. Study was only four weeks in duration, which is a snap-shot of a chronic life-long disease. Study was a single-center study which might not be a representative of the general population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes